CLINICAL TRIAL: NCT00470951
Title: A Comparison for Laparoscopically Assisted and Open Surgery for Advanced Rectal Cancer After Preoperative Chemoradiation- Randomized Prospective Trial
Brief Title: Randomized Prospective Trial for Laparoscopic vs Open Resection for Rectal Cancer
Acronym: CTS-179
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Seung Yong Jeong, Professor, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-179
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; laparoscopic assisted resection; open resection; preoperative chemoradiation; randomized trial
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- open rectal resection (Active Comparator): conventional open resection
  Interventions: Procedure: open rectal resection
- laparoscopic rectal resection (Active Comparator): laparoscopic rectal resection
  Interventions: Procedure: laparoscopic rectal resection

INTERVENTIONS:
Procedure: open rectal resection — open rectal resection
  Arms: open rectal resection
Procedure: laparoscopic rectal resection — laparoscopic assisted rectal resection
  Arms: laparoscopic rectal resection

SUMMARY:
The investigators designed the randomized prospective trial of comparing open and laparoscopic resection in locally advanced rectal cancer after preoperative chemoradiation in order to determine the oncologic and functional efficacy of laparoscopic rectal resection.

DETAILED DESCRIPTION:
1. Title: A comparison for laparoscopically assisted and open surgery for advanced rectal cancer after preoperative chemoradiation - randomized prospective trial
2. Principal investigator: Jae Hwan Oh Co-investigator: Seung Yong Jeong, Sung Bum Kang, Hyo Seong Choi, Seok-Byung Lim
3. Purpose of the study: To compare efficacy of laparoscopic and open resection for locally advanced rectal cancer after preoperative chemoradiation
4. Specific aims

   1. comparison of oncologic outcomes
   2. comparison of quality of life
   3. comparison of anorectal function
5. Materials Rectal cancer <9cm from anal verge, measured by rigid sigmoidoscopy histologically proven adenocarcinoma locally advanced (T3), determined by CT, transrectal ultrasonography, MRI without any contraindication for general anesthesia,operation and chemoradiation Completion of preoperative chemoradiation
6. Statistics

   1. Sample size calculation for non-inferiority trial: 340
   2. Disease free survival: Log-rank test,Cox regression analysis
   3. QOL and anorectal function: Repeated measured ANCOVA
7. Methods

   1. operation time of operation : 6-8 weeks after end of preoperative chemoradiation surgical technique standard total mesorectal excision and high ligation of inferior mesenteric vessels
   2. preoperative chemoradiation chemotherapy: 2 cycles of 5-FU (400 mg/m2/day) + LV (20 mg/m2/day) IV bolus, for 3 days in 1st & 5th wks of RT or Capecitabine 825 mg/m2 p.o. bid during RT RT:45 Gy/ 25 fractions to the pelvis, 5.4 Gy/ 3 fractions boost to the primary tumor over 5.5 wks
   3. postoperative chemotherapy 4 cycles of 5-FU (400 mg/m2/day) + LV (20 mg/m2/day) IV bolus, for 5 days, 4 wks interval
   4. oncologic outcomes

      1. Short-term outcomes Surgical length of incision op time blood loss intraoperative complications conversion rate Pathological resection margins (proximal, distal, circumferential) number of harvested lymph nodes length of resected bowel tumor regression grade (Dworak's grading) TNM staging Perioperative recovery duration of use of parenteral narcotics initiation of peristalsis initiation of oral intake duration of hospital stay 30-day postoperative mortality morbidity
      2. Long-term outcomes Primary end point Disease free survival (3 years after surgery) Secondary end points Overall survival Local recurrence Distant metastasis Port-site and wound site recurrence
   5. Quality of life Urinary function Duration of urinary catheterization Residual urine volume at discharge International Prostate Symptom Score (IPSS) Male sexual function International Index of Erectile Function (IIEF) Female sexual function Female Sexual Function Index (FSFI) QOL assessment EORTC QLQ C30 EORTC QLQ CR38
   6. Anorectal function Anorectal manometry Maximum Resting Pressure Maximum Squeezing Pressure High Pressure Zone Sphincter Length Sensory Threshold Rectal Capacity Rectal Compliance Rectoanal Inhibitory Reflex Fecal Incontinence Severity Index (FISI)

ELIGIBILITY:
Inclusion Criteria:

* Mid to low rectal cancer (within 9cm from AV, measured by RS)
* Histologically proven adenocarcinoma
* Locally advanced (T3, determined by CT, MRI and TRUS)
* Completion of preoperative chemoradiation
* Age: 18-80
* Hb ≥ 10g/dl, WBC≥ 3,000/mm3, Plt≥ 100,000/mm3
* Cr ≤ 1.5 mg/dl
* Adequate cardiopulmonary function
* Informed consent from patient or patient's relative

Exclusion Criteria:

* Metastasis in liver, lung, brain, bone, paraaortic LN, subclavicular LN, inguinal LN
* Second primary malignancy (except CIS of the cervix or adequately treated skin cancer or prior malignancy treated more than 5 years ago without recurrence)
* Cardiopulmonary dysfunction
* Active, uncontrolled infection
* Active, uncontrolled psychosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2006-04; Primary Completion 2012-08 (Actual); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 3 years

SECONDARY OUTCOMES:
Anorectal function | 1 year
Overall survival | 3 year, 5 year
Quality of life | preop, postop 3mo, posop 1 yr, 3yr, 5yr

OTHER OUTCOMES:
Immunologic response | preop, postop 2hr, postop 1day, 5day

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hwan Oh, M.D., ph.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Park JW, Kang SB, Hao J, Lim SB, Choi HS, Kim DW, Chang HJ, Kim DY, Jung KH, Kim TY, Kang GH, Chie EK, Kim SY, Sohn DK, Kim JS, Lee HS, Kim JH, Jeong SY, Oh JH. Open versus laparoscopic surgery for mid or low rectal cancer after neoadjuvant chemoradiotherapy (COREAN trial): 10-year follow-up of an open-label, non-inferiority, randomised controlled trial. Lancet Gastroenterol Hepatol. 2021 Jul;6(7):569-577. doi: 10.1016/S2468-1253(21)00094-7. Epub 2021 Apr 23. PMID 33894918
- [Derived] Park JS, Kang H, Park SY, Kim HJ, Woo IT, Park IK, Choi GS. Long-term oncologic after robotic versus laparoscopic right colectomy: a prospective randomized study. Surg Endosc. 2019 Sep;33(9):2975-2981. doi: 10.1007/s00464-018-6563-8. Epub 2018 Nov 19. PMID 30456502
- [Derived] Jeong SY, Park JW, Nam BH, Kim S, Kang SB, Lim SB, Choi HS, Kim DW, Chang HJ, Kim DY, Jung KH, Kim TY, Kang GH, Chie EK, Kim SY, Sohn DK, Kim DH, Kim JS, Lee HS, Kim JH, Oh JH. Open versus laparoscopic surgery for mid-rectal or low-rectal cancer after neoadjuvant chemoradiotherapy (COREAN trial): survival outcomes of an open-label, non-inferiority, randomised controlled trial. Lancet Oncol. 2014 Jun;15(7):767-74. doi: 10.1016/S1470-2045(14)70205-0. Epub 2014 May 15. PMID 24837215
- [Derived] Kang SB, Park JW, Jeong SY, Nam BH, Choi HS, Kim DW, Lim SB, Lee TG, Kim DY, Kim JS, Chang HJ, Lee HS, Kim SY, Jung KH, Hong YS, Kim JH, Sohn DK, Kim DH, Oh JH. Open versus laparoscopic surgery for mid or low rectal cancer after neoadjuvant chemoradiotherapy (COREAN trial): short-term outcomes of an open-label randomised controlled trial. Lancet Oncol. 2010 Jul;11(7):637-45. doi: 10.1016/S1470-2045(10)70131-5. Epub 2010 Jun 16. PMID 20610322